CLINICAL TRIAL: NCT00105872
Title: Behavioral Insomnia Therapy in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 00-091
Record Dates: First submitted 2005-03-17; First posted 2005-03-18 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-03

CONDITIONS: Insomnia; Primary Insomnia; Secondary Insomnia
Keywords: insomnia; cognitive behavior therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy

SUMMARY:
Insomnia reduces quality of life, increases risks for other illnesses, and enhances health care costs/utilization. Several efficacy studies have shown that Cognitive-Behavioral Therapy (CBT) for insomnia improves sleep and diurnal complaints among highly screened samples; however, its effectiveness among �real-world� primary care patients is yet to be tested. This project is highly relevant to the VA health care mission, given the high prevalence of insomnia in middle-aged and older adults. Pilot data from this VA suggest that 40% of primary care patients report trouble sleeping.

DETAILED DESCRIPTION:
Background:

Insomnia reduces quality of life, increases risks for other illnesses, and enhances health care costs/utilization. Several efficacy studies have shown that Cognitive-Behavioral Therapy (CBT) for insomnia improves sleep and diurnal complaints among highly screened samples; however, its effectiveness among �real-world� primary care patients is yet to be tested. This project is highly relevant to the VA health care mission, given the high prevalence of insomnia in middle-aged and older adults. Pilot data from this VA suggest that 40% of primary care patients report trouble sleeping.

Objectives:

This project tests the incremental benefits of adding CBT to usual primary care for reducing sleep disturbance, diurnal dysfunction, quality of life concerns and health care utilization among veterans enrolled in the DVAMC Primary Care Clinics. Study hypotheses predict that patients who receive CBT along with usual care will show greater improvements in sleep, mood, and quality of life, as well as larger reductions in health care utilization than will those who receive usual care alone.

Methods:

This is a single-blind, randomized, parallel group, clinical effectiveness study of 106 veteran insomnia sufferers. Eligibility criteria include: meeting structured interview criteria for insomnia, mean subjective total wake time of > 60 minutes per night, mental status score > 27 on Folstein MMSE, no unstable medical or psychiatric disorder, no polysomnographic evidence of sleep apnea or periodic limb movements, and approval of primary provider. Participants are randomly assigned to CBT + Usual Care or to Usual Care Control condition which provides therapist contact but no active behavioral treatment. Measures of sleep, mood, and quality of life are obtained before and after treatment and at a 6-month follow up. Computerized utilization data is obtained for the six months preceding and following treatment. A series of multivariate and univariate statistical tests will be conducted.

Status:

Major activities over the past year involved ongoing recruiting and enrolling participants. The study closed to enrollment on 7/19/05. Of 357 patients who completed screening procedures, 81 were eligible and enrolled in the project. Of these, five are in the pre-treatment phase, one is in the treatment phase, and 12 are in the post-treatment phase. Fifty-one patients have completed all study procedures. Eleven patients dropped out prior to completing the study, and one patient withdrew consent. A 1-year no cost extension was requested on 7/26/05 because of unavoidable delays in subject recruitment and enrollment, and we are awaiting a response.

ELIGIBILITY:
Inclusion Criteria:

1. Veteran enrolled in primary care at Durham VAMC
2. Insomnia complaint for > 1 month
3. Meet structured interview criteria for at least one DSM-IV insomnia subtype
4. Mean total wake time > 60 minutes per night
5. Provide informed consent
6. Concurrence for enrollment from primary care provider

Exclusion Criteria:

1. Terminal illness
2. Acute or unstable psychiatric condition
3. Acute pain or poorly managed chronic pain
4. Not mentally competent
5. Evidence of clinically significant sleep apnea or periodic limb movement disorder
6. Refuse to provide informed consent
7. In the opinion of their MD provider, have an unstable psychiatric or medical condition that makes participation unadvisable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-03; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Objective (actigraphic) and subjective (sleep log) sleep measures at 6 weeks and 6 months

SECONDARY OUTCOMES:
Mood and quality of life at 6 weeks and 6 months; healthcare utilization at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jack D. Edinger, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Edinger JD, Glenn DM, Bastian LA, Marsh GR, Dailey D, Hope TV, Young M, Shaw E, Meeks G. Daytime testing after laboratory or home-based polysomnography: comparisons of middle-aged insomnia sufferers and normal sleepers. J Sleep Res. 2003 Mar;12(1):43-52. doi: 10.1046/j.1365-2869.2003.00335.x. PMID 12603786
- [Result] Edinger JD, Means MK, Stechuchak KM, Olsen MK. A pilot study of inexpensive sleep-assessment devices. Behav Sleep Med. 2004;2(1):41-9. doi: 10.1207/s15402010bsm0201_4. PMID 15600223
- [Result] Edinger JD, Olsen MK, Stechuchak KM, Means MK, Lineberger MD, Kirby A, Carney CE. Cognitive behavioral therapy for patients with primary insomnia or insomnia associated predominantly with mixed psychiatric disorders: a randomized clinical trial. Sleep. 2009 Apr;32(4):499-510. doi: 10.1093/sleep/32.4.499. PMID 19413144